CLINICAL TRIAL: NCT01345682
Title: A Randomised, Open-label, Phase III Study to Evaluate the Efficacy and Safety of Oral Afatinib (BIBW 2992) Versus Intravenous Methotrexate in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma Who Have Progressed After Platinum-based Therapy
Brief Title: LUX-Head&Neck 1: A Phase III Trial of Afatinib (BIBW2992) Versus Methotrexate for the Treatment of Recurrent and/or Metastatic (R/M) Head and Neck Squamous Cell Cancer After Platinum Based Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.43; 2011-000391-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Afatinib; Methotrexate

ARMS (2):
- Afatinib (BIBW 2992) (Experimental): Once daily
  Interventions: Drug: Afatinib
- Methotrexate (Active Comparator): Weekly
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Afatinib — Once daily
  Arms: Afatinib (BIBW 2992)
Drug: Methotrexate — Weekly
  Arms: Methotrexate

SUMMARY:
This randomised, open-label, phase III study will be performed in patients with R/M head and neck squamous cell carcinoma (HNSCC) who have progressed after platinum-based therapy. The objectives of the trial are to compare the efficacy and safety of afatinib versus methotrexate

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically confirmed R/M HNSCC of the oral cavity, oropharynx, hypopharynx or larynx, not amenable for salvage surgery or radiotherapy
2. Documented progressive disease based on investigator assessment according to Response Evaluation Criteria in Solid Tumours (RECIST) following receipt of at least two cycles of cisplatin or carboplatin administered for R/M disease
3. Measurable disease according to RECIST
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion criteria:

1. Progressive disease within three months of completion of curatively intended treatment for locoregionally advanced or metastatic HNSCC
2. Any other than one previous platinum based systemic regimen given for R/M disease
3. Prior treatment with epidermal growth factor receptor (EGFR)-targeted small molecules
4. Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2014-03-15 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (101):
- United States (8):
  - 1200.43.00113 Boehringer Ingelheim Investigational Site, Harvey, Illinois
  - 1200.43.00106 Boehringer Ingelheim Investigational Site, Peoria, Illinois
  - 1200.43.00110 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1200.43.00107 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1200.43.00105 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 1200.43.00102 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1200.43.00103 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1200.43.00109 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Argentina (3):
  - 1200.43.05401 Boehringer Ingelheim Investigational Site, Ciudad Autonoma de Bs As
  - 1200.43.05402 Boehringer Ingelheim Investigational Site, Santa Fe
  - 1200.43.05403 Boehringer Ingelheim Investigational Site, Villa Domínico
- Austria (3):
  - 1200.43.04303 Boehringer Ingelheim Investigational Site, Leoben
  - 1200.43.04305 Boehringer Ingelheim Investigational Site, Salzburg
  - 1200.43.04301 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (4):
  - 1200.43.03202 Boehringer Ingelheim Investigational Site, Brussels
  - 1200.43.03203 Boehringer Ingelheim Investigational Site, Edegem
  - 1200.43.03204 Boehringer Ingelheim Investigational Site, Ghent
  - 1200.43.03201 Boehringer Ingelheim Investigational Site, Leuven
- Brazil (7):
  - 1200.43.05504 Boehringer Ingelheim Investigational Site, Barretos
  - 1200.43.05505 Boehringer Ingelheim Investigational Site, Jaú
  - 1200.43.05507 Boehringer Ingelheim Investigational Site, Passo Fundo
  - 1200.43.05503 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1200.43.05502 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 1200.43.05501 Boehringer Ingelheim Investigational Site, São Paulo
  - 1200.43.05506 Boehringer Ingelheim Investigational Site, São Paulo
- Czechia (3):
  - 1200.43.04202 Boehringer Ingelheim Investigational Site, Olomouc
  - 1200.43.04201 Boehringer Ingelheim Investigational Site, Prague
  - 1200.43.04203 Boehringer Ingelheim Investigational Site, Prague
- 1200.43.04501 Boehringer Ingelheim Investigational Site, København Ø, Denmark
- France (13):
  - 1200.43.03304 Boehringer Ingelheim Investigational Site, Avignon
  - 1200.43.03306 Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1200.43.03312 Boehringer Ingelheim Investigational Site, Dijon
  - 1200.43.03303 Boehringer Ingelheim Investigational Site, Lille
  - 1200.43.03301 Boehringer Ingelheim Investigational Site, Lyon
  - 1200.43.03302 Boehringer Ingelheim Investigational Site, Montpellier
  - 1200.43.03307 Boehringer Ingelheim Investigational Site, Nice
  - 1200.43.03314 Boehringer Ingelheim Investigational Site, Paris
  - 1200.43.03305 Boehringer Ingelheim Investigational Site, Poitiers
  - 1200.43.03316 Boehringer Ingelheim Investigational Site, Rouen
  - 1200.43.03309 Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1200.43.03310 Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
  - 1200.43.03317 Boehringer Ingelheim Investigational Site, Villejuif
- Germany (9):
  - 1200.43.04903 Boehringer Ingelheim Investigational Site, Aachen
  - 1200.43.04902 Boehringer Ingelheim Investigational Site, Berlin
  - 1200.43.04909 Boehringer Ingelheim Investigational Site, Dresden
  - 1200.43.04901 Boehringer Ingelheim Investigational Site, Essen
  - 1200.43.04905 Boehringer Ingelheim Investigational Site, Hamburg
  - 1200.43.04906 Boehringer Ingelheim Investigational Site, Hanover
  - 1200.43.04908 Boehringer Ingelheim Investigational Site, Jena
  - 1200.43.04904 Boehringer Ingelheim Investigational Site, Leipzig
  - 1200.43.04907 Boehringer Ingelheim Investigational Site, Mannheim
- Greece (3):
  - 1200.43.03004 Boehringer Ingelheim Investigational Site, Haidari
  - 1200.43.03005 Boehringer Ingelheim Investigational Site, Heraklion
  - 1200.43.03002 Boehringer Ingelheim Investigational Site, Thessaloniki
- Israel (3):
  - 1200.43.97201 Boehringer Ingelheim Investigational Site, Haifa
  - 1200.43.97203 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1200.43.97204 Boehringer Ingelheim Investigational Site, Tel Litwinsky
- Italy (10):
  - 1200.43.03909 Boehringer Ingelheim Investigational Site, Aosta
  - 1200.43.03908 Boehringer Ingelheim Investigational Site, Cagliari
  - 1200.43.03901 Boehringer Ingelheim Investigational Site, Confreria (CN)
  - 1200.43.03907 Boehringer Ingelheim Investigational Site, Milan
  - 1200.43.03903 Boehringer Ingelheim Investigational Site, Napoli
  - 1200.43.03905 Boehringer Ingelheim Investigational Site, Palermo
  - 1200.43.03902 Boehringer Ingelheim Investigational Site, Savona
  - 1200.43.03904 Boehringer Ingelheim Investigational Site, Taormina (ME)
  - 1200.43.03906 Boehringer Ingelheim Investigational Site, Venezia
  - 1200.43.03910 Boehringer Ingelheim Investigational Site, Viterbo
- Japan (13):
  - 1200.43.08106 Boehringer Ingelheim Investigational Site, Aichi, Nagoya
  - 1200.43.08103 Boehringer Ingelheim Investigational Site, Chiba, Kashiwa
  - 1200.43.08108 Boehringer Ingelheim Investigational Site, Ehime, Matsuyama
  - 1200.43.08111 Boehringer Ingelheim Investigational Site, Hyogo, Akashi
  - 1200.43.08107 Boehringer Ingelheim Investigational Site, Hyogo, Kobe
  - 1200.43.08109 Boehringer Ingelheim Investigational Site, Kanagawa, Isehara
  - 1200.43.08114 Boehringer Ingelheim Investigational Site, Miyagi, Natori
  - 1200.43.08110 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1200.43.08105 Boehringer Ingelheim Investigational Site, Shizuoka, Sunto-gun
  - 1200.43.08102 Boehringer Ingelheim Investigational Site, Tochigi, Shimotsuke
  - 1200.43.08113 Boehringer Ingelheim Investigational Site, Tokyo, Koto-ku
  - 1200.43.08104 Boehringer Ingelheim Investigational Site, Tokyo, Meguro-ku
  - 1200.43.08112 Boehringer Ingelheim Investigational Site, Tokyo, Minato-ku
- 1200.43.05202 Boehringer Ingelheim Investigational Site, México, Mexico
- Russia (7):
  - 1200.43.00704 Boehringer Ingelheim Investigational Site, Ivanovo
  - 1200.43.00706 Boehringer Ingelheim Investigational Site, Kurski
  - 1200.43.00709 Boehringer Ingelheim Investigational Site, Moscow
  - 1200.43.00703 Boehringer Ingelheim Investigational Site, Omsk
  - 1200.43.00710 Boehringer Ingelheim Investigational Site, Pyatigorsk
  - 1200.43.00707 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1200.43.00705 Boehringer Ingelheim Investigational Site, Ufa
- South Africa (4):
  - 1200.43.02703 Boehringer Ingelheim Investigational Site, Cape Town
  - 1200.43.02704 Boehringer Ingelheim Investigational Site, Kraaifontein, Cape Town
  - 1200.43.02701 Boehringer Ingelheim Investigational Site, Parktown, Johannesburg
  - 1200.43.02702 Boehringer Ingelheim Investigational Site, Pretoria
- Spain (6):
  - 1200.43.03401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.43.03404 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.43.03405 Boehringer Ingelheim Investigational Site, Girona
  - 1200.43.03406 Boehringer Ingelheim Investigational Site, Málaga
  - 1200.43.03402 Boehringer Ingelheim Investigational Site, Salamanca
  - 1200.43.03403 Boehringer Ingelheim Investigational Site, Zaragoza
- 1200.43.04602 Boehringer Ingelheim Investigational Site, Gothenburg, Sweden
- Switzerland (2):
  - 1200.43.04101 Boehringer Ingelheim Investigational Site, Basel
  - 1200.43.04102 Boehringer Ingelheim Investigational Site, Bern

REFERENCES:
- [Derived] Cohen EEW, Licitra LF, Burtness B, Fayette J, Gauler T, Clement PM, Grau JJ, Del Campo JM, Mailliez A, Haddad RI, Vermorken JB, Tahara M, Guigay J, Geoffrois L, Merlano MC, Dupuis N, Kramer N, Cong XJ, Gibson N, Solca F, Ehrnrooth E, Machiels JH. Biomarkers predict enhanced clinical outcomes with afatinib versus methotrexate in patients with second-line recurrent and/or metastatic head and neck cancer. Ann Oncol. 2017 Oct 1;28(10):2526-2532. doi: 10.1093/annonc/mdx344. PMID 28961833
- [Derived] Clement PM, Gauler T, Machiels JP, Haddad RI, Fayette J, Licitra LF, Tahara M, Cohen EE, Cupissol D, Grau JJ, Guigay J, Caponigro F, de Castro G Jr, de Souza Viana L, Keilholz U, Del Campo JM, Cong XJ, Ehrnrooth E, Vermorken JB; LUX-H&N 1 investigators. Afatinib versus methotrexate in older patients with second-line recurrent and/or metastatic head and neck squamous cell carcinoma: subgroup analysis of the LUX-Head & Neck 1 trial. Ann Oncol. 2016 Aug;27(8):1585-93. doi: 10.1093/annonc/mdw151. Epub 2016 Apr 15. PMID 27084954
- [Derived] Machiels JP, Haddad RI, Fayette J, Licitra LF, Tahara M, Vermorken JB, Clement PM, Gauler T, Cupissol D, Grau JJ, Guigay J, Caponigro F, de Castro G Jr, de Souza Viana L, Keilholz U, Del Campo JM, Cong XJ, Ehrnrooth E, Cohen EE; LUX-H&N 1 investigators. Afatinib versus methotrexate as second-line treatment in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 1): an open-label, randomised phase 3 trial. Lancet Oncol. 2015 May;16(5):583-94. doi: 10.1016/S1470-2045(15)70124-5. Epub 2015 Apr 16. PMID 25892145

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib (BIBW 2992): Oral administration of Afatinib (film-coated tablets). Starting dose 40 milligram (mg) once daily; escalation to 50 mg/day and / or dose reduction to 40 mg/day (if applicable), 30 mg/day, or 20 mg/day (according to the protocol-defined dose escalation and dose reduction scheme) if required. No dose increase was allowed after a dose reduction.
- Methotrexate: Intravenous bolus injection of Methotrexate Starting dose 40 mg/m² weekly; escalation to 50 mg/m² and / or dose reduction to 40 mg/m² (if applicable), 30 mg/m², and 20 mg/m² (according to the protocol-defined dose escalation and dose reduction scheme) if required. No dose increase was allowed after a dose reduction.
Period: Overall Study
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Started | 322 (Randomised) | 161 (Randomised)
Completed | 0 | 0
Not Completed | 322 | 161
Not completed — Progressive disease per RECIST | 226 | 93
Not completed — Worsening of underlying cancer disease | 23 | 12
Not completed — Adverse Event | 51 | 41
Not completed — Non-compliance with protocol | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Refused to continue trial medication | 16 | 9
Not completed — Not treated | 2 | 1
Not completed — Reason other than those specified above | 4 | 3

BASELINE CHARACTERISTICS:
Population: The randomised set (RS) included all patients who were randomised to receive treatment, whether treated or not
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib (BIBW 2992) | Methotrexate | Total
Number analyzed (Participants) | 322 | 161 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (8.8) | 59.3 (9.7) | 59.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 24 | 71
  Male | 275 | 137 | 412

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Central Independent Review
Description: PFS was defined as the time from the date of randomisation to disease progression or death, whichever occurred first. The primary analysis of PFS considered PFS events as assessed by central independent review, including all data collected until the study completion date (06 December 2016).
  The date of disease progression was recorded based on RECIST version 1.1. Unequivocal progression of disease was determined if at least one of the following criteria applied:
  * At least 20% increase in the Sum of Diameters (SoD) of target lesions taking as reference the smallest SoD recorded since the treatment started, together with an absolute increase in the SoD of at least 5 mm
  * Appearance of one or more new lesions
  * Unequivocal progression of existing non-target lesions
Time Frame: From randomization until disease progression, death or study completion date (06Dec2016); Up to 60 months
Population: Randomised set (RS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 322 | 161
months | 2.63 [2.10 to 2.73] | 1.74 [1.48 to 2.40]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.0257, Stratified Log-rank test — Log-rank test stratified by baseline Eastern Cooperative Oncology Group (ECOG) Performance score (PS)(0 or 1) and prior use of Epidermal Growth Factor Receptor (EGFR)-targeted antibody in the Recurrent and/or Metastatic (R/M) setting (Yes or No); Hazard Ratio (HR) = 0.792, 95% CI 2-sided [0.643 to 0.977] — Hazard ratio from Cox proportional hazards model stratified by baseline ECOG PS (0 or 1) and prior use of EGFR-targeted antibody in the R/M setting (Yes or No). Afatinib (BIBW 2992) vs Methotrexate

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was a key secondary endpoint of this trial. OS was defined as the time from randomisation to death (irrespective of the cause of death). Patients for whom there was no evidence of death at the study completion date (06 December 2016) were to be censored on the date that they were last known to be alive.
Time Frame: From randomization until death or study completion date (06Dec2016); Up to 60 months
Population: RS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 322 | 161
months | 6.87 [6.14 to 7.79] | 6.01 [5.16 to 7.75]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.6755, Stratified Log-rank test — Log-rank test stratified by baseline ECOG PS (0 or 1) and prior use of EGFR-targeted antibody in the R/M setting (Yes or No); Hazard Ratio (HR) = 0.958, 95% CI 2-sided [0.786 to 1.169] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response (OR)
Description: OR is defined as the best overall response of complete response (CR) and partial response (PR) according to RECIST version 1.1, CR for target lesions (TL): Disappearance of all target lesions. CR for non-target lesions (NTL): Disappearance of all non-target lesions. All lymph nodes must be non-pathological in size (<10mm short axis).
  PR for TL: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
  Other factors which add to the overall response of an imaging timepoint as PR are as below:-
  * CR in TL, but non-CR/Non-Progressive Disease (PD) in NTL leads to PR
  * CR in TL, but not evaluated NTL leads to PR
  * PR in TL, but non-PD NTL or not all evaluated NTL leads to PR;
  All the above scenarios should also satisfy 'No occurrence of new lesions'.
Time Frame: Tumour imaging was to be performed every 6 weeks during the first 24 weeks of treatment, and hereafter every 8 weeks (data cut-off 07May2014); Up to 28 months
Population: RS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 322 | 161
percentage of participants | 10.2 [7.16 to 14.09] | 5.6 [2.58 to 10.34]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.1010, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.88 to 4.14] — Odds ratio, 95% Confidence Interval (CI) and p-value (two-sided) from logistic regression stratified by baseline ECOG PS (0 or 1) and prior use of EGFR-targeted antibody in the R/M setting (Yes or No). Afatinib (BIBW 2992) vs Methotrexate

4. Secondary Outcome: Disease Control (DC)
Description: DC is defined as the best overall response of CR, PR, stable disease (SD) and non-CR/non-PD.
  CR for target lesions (TL): Disappearance of all target lesions. CR for non-target lesions (NTL): Disappearance of all non-target lesions . All lymph nodes must be non-pathological in size (<10mm short axis).
  PR for TL: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
  Other factors which add to the overall response of an imaging timepoint as PR are as below:-
  * CR in TL, but non-CR/Non-PD in NTL leads to PR
  * CR in TL, but not evaluated NTL leads to PR
  * PR in TL, but non-PD NTL or not all evaluated NTL leads to PR;
  SD for TL: change in the sum of diameters does not satisfy PR or PD.
  SD in TL, non-PD in NTL lead to overall response of SD, provided there is no appearance of new lesions.
Time Frame: as for outcome 3
Population: RS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 322 | 161
percentage of participants | 49.1 [43.48 to 54.67] | 38.5 [30.95 to 46.49]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.0353, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.03 to 2.26] — Odds ratio, 95% CI and p-value (two-sided) from logistic regression stratified by baseline ECOG PS (0 or 1) and prior use of EGFR-targeted antibody in the R/M setting (Yes or No). Afatinib (BIBW 2992) vs Methotrexate

5. Secondary Outcome: Tumour Shrinkage
Description: Tumour shrinkage, defined as the maximum decrease from baseline in the sum of diameters of the target lesions, as measured by central imaging. The longest diameter of target lesions was recorded, except for lymph nodes, which were measured by their short axis.
  Negative values indicate a reduction in the sum of target lesion diameters and positive values an increase.
  Percentage of Participants with Tumour shrinkage as per the categories (>=20% increase, >=0 - <20% increase, >0 - <30% decrease, >=30 - <50% decrease, >=50% decrease) are presented.
Time Frame: as for outcome 3
Population: RS (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 248 | 121
percentage of participants
  >=20% increase | 16.5 | 21.1
  >=0 - <20% increase | 24.2 | 31.1
  >0 - <30% decrease | 23.6 | 16.1
  >=30 - <50% decrease | 6.2 | 4.3
  >=50% decrease | 5.0 | 1.9

6. Secondary Outcome: Health Related Quality of Life (HRQOL)- Change in Pain Scores Over Time
Description: The HRQOL analyses focused on pain, swallowing, and global health status measured by the European Organisation for Research and Treatment of Cancer [EORTC] quality of life questionnaires Core 30 [QLQ-C30], and head and neck cancer specific supplementary module EORTC QLQ-H&N35:
  Pain scale from H&N35, Swallowing scale from H&N35 and Global health status/QoL scale from C30.
  Pain scale includes items 31-34 from H&N 35; Swallowing scale includes items 35-38 from H&N35 and Global health status/QoL scale includes items 29-30 from C30.
  The scores of these scales were averaged from the scores of the component items, transformed and analyzed on 0 - 100 scale. For pain and swallowing scales, higher scores represent worse outcome; for the global health/QoL scale, higher scores represent better outcome.
  Changes in scores over time were assessed using longitudinal models.
  The analyses of HRQOL are presented for the 07 May 2014 cut-off date.
Time Frame: From randomization until one month after discontinuation of study medication, death or data cut-off (07May2014); Up to 28 months.
Population: RS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 265 | 117
scores on a scale | 11.8 (3.16) | 16.2 (3.43)
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Changes in scores over time were assessed using longitudinal models, i.e. mixed effects growth curve models with the average profile over time for each endpoint described by a piecewise linear model adjusted for the fixed effects baseline ECOG performance score (PS) and prior use of EGFR-targeted antibody for recurrent and/or metastatic head and neck squamous cell carcinoma (R/M HNSCC); Test type: Superiority or Other; p = 0.0300, longitudinal models — Adjusted for baseline ECOG performance score (0 or 1) and prior use of EGFR-targeted antibody for R/M HNSCC (Yes or No); Adjusted mean difference = -4.4, 95% CI 2-sided [-8.31 to -0.42], Standard Error of Mean 2.01 — Afatinib (BIBW 2992) vs Methotrexate

7. Secondary Outcome: Health Related Quality of Life (HRQOL)- Change in Swallowing Scores Over Time
Description: as for outcome 6
Time Frame: as for outcome 6
Population: RS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 257 | 112
scores on a scale | 20.0 (3.40) | 20.1 (3.66)
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Changes in scores over time were assessed using longitudinal models, i.e. mixed effects growth curve models with the average profile over time for each endpoint described by a piecewise linear model adjusted for the fixed effects baseline ECOG PS and prior use of EGFR-targeted antibody for recurrent and/or metastatic head and neck squamous cell carcinoma (R/M HNSCC); Test type: Superiority or Other; p = 0.9773, longitudinal models — Adjusted for baseline ECOG performance score (0 or 1) and prior use of EGFR-targeted antibody for R/M HNSCC (Yes or No); Adjusted mean difference = -0.1, 95% CI 2-sided [-4.30 to 4.18], Standard Error of Mean 2.16 — Afatinib (BIBW 2992) vs Methotrexate

8. Secondary Outcome: Health Related Quality of Life (HRQOL)- Change in Global Health Scores Over Time
Description: as for outcome 6
Time Frame: as for outcome 6
Population: RS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 267 | 117
scores on a scale | 28.7 (3.54) | 28.2 (3.76)
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.7767, longitudinal models — Adjusted for baseline ECOG performance score (0 or 1) and prior use of EGFR-targeted antibody for R/M HNSCC (Yes or No); Adjusted mean difference = 0.6, 95% CI 2-sided [-3.28 to 4.39], Standard Error of Mean 1.95 — Afatinib (BIBW 2992) vs Methotrexate

9. Secondary Outcome: Status Change in Pain Scale
Description: Distribution of patients with improved, stable or worsened HRQOL: Improvement was defined as a score improved by at least 10 points from baseline (on the 0-100 point scale) at any time during the trial. If a patient had not improved, worsening was defined as a 10-point worsening at any time during the trial. Otherwise, a patient was considered as stable.
Time Frame: as for outcome 6
Population: RS (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 265 | 117
percentage of participants
  Improved | 26.4 | 23.1
  Stable | 32.1 | 31.6
  Worsened | 41.5 | 45.3
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.494, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.717 to 1.990] — [estimate comment as in outcome 4, analysis 1]

10. Secondary Outcome: Status Change in Swallowing Scale
Description: as for outcome 9
Time Frame: as for outcome 6
Population: RS (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 257 | 112
percentage of participants
  Improved | 26.1 | 23.2
  Stable | 34.2 | 29.5
  Worsened | 39.7 | 47.3
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.584, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.687 to 1.950] — [estimate comment as in outcome 4, analysis 1]

11. Secondary Outcome: Status Change in Global Health Status Scale
Description: as for outcome 9
Time Frame: as for outcome 6
Population: RS (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 267 | 117
percentage of participants
  Improved | 30.3 | 29.1
  Stable | 26.6 | 25.6
  Worsened | 43.1 | 45.3
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.816, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.657 to 1.705] — [estimate comment as in outcome 4, analysis 1]

12. Secondary Outcome: Time to Deterioration in Pain
Description: The time to deterioration was defined as the time from randomisation to a score increased (i.e. worsened) by at least 10 points from baseline (0-100 point scale). If score is missing, and patient died within 28 days after scheduled time for completion, the patient was considered deteriorated. In this case, time to deterioration is time to death.
Time Frame: as for outcome 6
Population: RS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 322 | 161
months | 3.02 [2.83 to 3.75] | 2.30 [1.64 to 3.32]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.0217, Stratified Log-rank test — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.55 to 0.96] — Hazard ratio from Cox proportional hazards model stratified by baseline ECOG PS (0 or 1) and prior use of EGFR-targeted antibody in the R/M setting (Yes or No)

13. Secondary Outcome: Time to Deterioration in Swallowing
Description: as for outcome 12
Time Frame: as for outcome 6
Population: RS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 322 | 161
months | 3.75 [2.83 to 4.30] | 2.10 [1.48 to 3.32]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.0040, Stratified Log-rank test — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.50 to 0.89] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Time to Deterioration in Global Health Status
Description: The time to deterioration was defined as the time from randomisation to a score decreased (i.e. worsened) by at least 10 points from baseline (0-100 point scale). If score is missing, and patient died within 28 days after scheduled time for completion, the patient was considered deteriorated. In this case, time to deterioration is time to death.
Time Frame: as for outcome 6
Population: RS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Number analyzed (Participants) | 322 | 161
months | 3.25 [2.83 to 4.01] | 2.69 [1.61 to 2.86]
Statistical Analysis 1: Comparison: Afatinib (BIBW 2992) vs Methotrexate; Test type: Superiority or Other; p = 0.0268, Stratified Log-rank test — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.56 to 0.97] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first administration of study medication (afatinib or methotrexate) and within 28 days after the last administration of study medication (study completion date is 06Dec2016); Up to 60 months
Groups:
- Methotrexate: Intravenous bolus injection of Methotrexate Starting dose 40 milligram per square meter mg/m² weekly; escalation to 50 mg/m² and / or dose reduction to 40 mg/m² (if applicable), 30 mg/m², and 20 mg/m² (according to the protocol-defined dose escalation and dose reduction scheme) if required. No dose increase was allowed after a dose reduction.
Arm/Group | Afatinib (BIBW 2992) | Methotrexate
Serious Adverse Events (participants affected / at risk) | 168/320 | 73/160
Other Adverse Events (participants affected / at risk) | 309/320 | 146/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (BIBW 2992) (N=320) | Methotrexate (N=160)
Anaemia (Blood and lymphatic system disorders) | 3 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 3 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 9 | 3
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Odynophagia (Gastrointestinal disorders) | 2 | 0
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 10 | 1
Asthenia (General disorders) | 6 | 1
Complication associated with device (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Face oedema (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 2
General physical health deterioration (General disorders) | 27 | 8
Hyperpyrexia (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Mucosal haemorrhage (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 3 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 7 | 5
Sudden death (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 4 | 0
Empyema (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 4 | 2
Oral infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 13 | 3
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 | 1
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Blood pressure orthostatic decreased (Investigations) | 1 | 0
False positive investigation result (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1
Dehydration (Metabolism and nutrition disorders) | 9 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Food aversion (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 1
Malnutrition (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 40 | 9
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 5 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Device dislocation (Product Issues) | 0 | 1
Device leakage (Product Issues) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Renal failure (Renal and urinary disorders) | 6 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrostomy (Surgical and medical procedures) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 4
Hypotension (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (BIBW 2992) (N=320) | Methotrexate (N=160)
Anaemia (Blood and lymphatic system disorders) | 61 | 42
Leukopenia (Blood and lymphatic system disorders) | 3 | 13
Neutropenia (Blood and lymphatic system disorders) | 1 | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 10
Abdominal pain (Gastrointestinal disorders) | 27 | 5
Constipation (Gastrointestinal disorders) | 39 | 28
Diarrhoea (Gastrointestinal disorders) | 239 | 28
Dyspepsia (Gastrointestinal disorders) | 31 | 4
Dysphagia (Gastrointestinal disorders) | 42 | 12
Nausea (Gastrointestinal disorders) | 89 | 43
Stomatitis (Gastrointestinal disorders) | 73 | 28
Vomiting (Gastrointestinal disorders) | 63 | 26
Asthenia (General disorders) | 66 | 41
Fatigue (General disorders) | 72 | 42
Mucosal inflammation (General disorders) | 74 | 42
Pyrexia (General disorders) | 38 | 27
Conjunctivitis (Infections and infestations) | 25 | 4
Folliculitis (Infections and infestations) | 24 | 1
Paronychia (Infections and infestations) | 51 | 0
Alanine aminotransferase increased (Investigations) | 4 | 19
Aspartate aminotransferase increased (Investigations) | 6 | 20
Weight decreased (Investigations) | 69 | 25
Decreased appetite (Metabolism and nutrition disorders) | 60 | 39
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 17 | 9
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 | 9
Headache (Nervous system disorders) | 26 | 16
Anxiety (Psychiatric disorders) | 21 | 7
Insomnia (Psychiatric disorders) | 27 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 | 5
Acne (Skin and subcutaneous tissue disorders) | 28 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 68 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 47 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 1
Rash (Skin and subcutaneous tissue disorders) | 134 | 11
Skin fissures (Skin and subcutaneous tissue disorders) | 40 | 0
Hypotension (Vascular disorders) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.